CLINICAL TRIAL: NCT04609839
Title: TeleRea'nCo : FOLLOW-UP OF PATIENTS WITH COVID-19.
Brief Title: FOLLOW-UP OF PATIENTS WITH COVID-19.
Acronym: TeleRea'nCo
Status: Withdrawn | Type: Observational
Why Stopped: Patients were enrolled in another similar clinical study
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: TeleRea'nCo; 7883 (Other: Hôpitaux Universitaires de Strasborug)
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Patient Admitted to Intensive Care Unit for COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient admitted to intensive care unit for COVID-19
  Interventions: Other: Follow-up of patients with COVID-19

INTERVENTIONS:
Other: Follow-up of patients with COVID-19 — The presence of sequelae, number of re-hospitalizations, date of death and cost of health expenditure will be collected.
  The Quality of life score (SF-36 questionnaire) and the Pittsburgh sleep quality index (PSQI questionnaire) will be completed by patients.

SUMMARY:
Some patients admitted to intensive care for a severe form of COVID-19 could have respiratory, cardiac, renal and neurological sequelae in the medium or long term.

The results of this research will allow an improvement in the understanding and management of patients in the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to intensive care unit for COVID-19
* Adult patient ≥ 18 years old
* Subject having expressed his non-opposition to the research
* Subject affiliated to a social health insurance protection scheme or beneficiary of such a scheme

Exclusion Criteria:

* Subject under safeguard of justice
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to intensive care unit for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
The presence of respiratory, renal, cardiac, motor, neurological, and psychological sequelae will be assessed by specialist doctors during the 12 months following the patient's discharge from intensive care. | The primary endpoint will be measured during 12 months following the patient's discharge from intensive care.

SECONDARY OUTCOMES:
1) The sequelae by type of impairment will be assessed by specialist doctors at 3, 6 and 12 months | At M3 (+/-15 days) : 3 months after patient inclusion-At M6 (+/-15 days) : 6 months after patient inclusion-At M12 (+/-15 days) : 12 months after patient inclusion
2) Number of re-hospitalizations at 3, 6 and 12 months | At M3 (+/-15 days) : 3 months after patient inclusion-At M6 (+/-15 days) : 6 months after patient inclusion-At M12 (+/-15 days) : 12 months after patient inclusion
3) Date of death | Date of death will be collected from inclusion to M12 (12 months after patient inclusion)
4.1) Quality of life score (SF-36 questionnaire) at 3, 6 and 12 months | At M3 (+/-15 days) : 3 months after patient inclusion-At M6 (+/-15 days) : 6 months after patient inclusion-At M12 (+/-15 days) : 12 months after patient inclusion
4.2) The Pittsburgh sleep quality index (PSQI questionnaire) at 3, 6 and 12 months | At M3 (+/-15 days) : 3 months after patient inclusion-At M6 (+/-15 days) : 6 months after patient inclusion-At M12 (+/-15 days) : 12 months after patient inclusion
5) Cost of health expenditure | The cost of health expenditure will be collected from inclusion to M12 (12 months after patient inclusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No